CLINICAL TRIAL: NCT06108193
Title: A Phase I/II Clinical Study of Topical Minoxidil in Acne Vulgaris
Brief Title: Toxicity and Efficacy Evaluation of Topical Minoxidil in Acne Vulgaris
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Lung Hsu, Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202001720A0
Record Dates: First submitted 2023-06-08; First posted 2023-10-30 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Acne Vulgaris
Keywords: androgen receptor; minoxidil
MeSH Terms: conditions — Acne Vulgaris; Bulbo-Spinal Atrophy, X-Linked | interventions — Minoxidil

STUDY DESIGN:
Intervention Model Description: PBF Minoxidil Solution 5% PBF Minoxidil Solution 2% Split face: 2% or 5% topical minoxidil solution applied and no treatment Description: Subjects will apply the 2% or 5% topical minoxidil solution to every inflammatory acne facial lesion on one half of the face and no treatment to every inflammatory acne lesion on the other half of the face twice a day for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- topical minoxidil in Acne Vulgaris (Experimental): Split face: 2% or 5% topical minoxidil solution applied and no treatment Description: Subjects will apply the 2% or 5% topical minoxidil solution to every inflammatory acne facial lesion on one half of the face and no treatment to every inflammatory acne lesion on the other half of the face twice a day for 4 weeks.
  Interventions: Drug: topical minoxidil in Acne Vulgaris

INTERVENTIONS:
Drug: topical minoxidil in Acne Vulgaris — Split face: 2% or 5% topical minoxidil solution applied and no treatment Description: Subjects will apply the 2% or 5% topical minoxidil solution to every inflammatory acne facial lesion on one half of the face and no treatment to every inflammatory acne lesion on the other half of the face twice a day for 4 weeks.

SUMMARY:
Patients with acne vulgaris (AV) appeared to be a chronic inflammation with a wide range in teenagers and adult. The protocol design is as follows.

The subjects enrolled through inclusion and exclusion criteria will undergo the blood and urine biochemical tests for baseline record. The photos from the subjects will be recorded per day, and the blood and urine biochemical tests will be recorded per week.

Objectives: primary: to test the toxicity of topical minoxidil in treatment of acne vulgaris; second: to evaluate the response and disease control rate in this pilot study.

Measurement: Time to resolution of individual acne lesions (14 days) Monitor of treatment efficacy: number of inflammatory acne lesions counting, time to resolution of individual acne lesion, and degree of acne severity measurement.

DETAILED DESCRIPTION:
1. Background 1.1 Overview of disease pathogenesis, epidemiology and current treatments Patients with acne vulgaris (AV) appeared to be a chronic inflammation with a wide range in teenagers and adult. There are four main components in the pathogenesis of AV: (1) enhancement of sebum secretion (2) keratinization of the middle infundibulum (3) bacterial proliferation of the follicle (4) Inflammation. In sebaceous glands, pro-hormones dehydroepiandrosterone (DHEA) and androstenedione can be metabolized into testosterone and dehydrotestosterone (DHT). Literature identified androgen receptor (AR) expression in sebaceous glands by immunohistochemistry and high sebum secretion associated with high AR expression in sebaceous gland of T-zone than U-zone of face. Via AR, androgen could induce sebocyte sebaceous differentiation. Genomic related studies elucidated AR related genes were associated with severe acne. Imbalanced androgen correlated with AR plays an important role in increasing sebaceous glands excretion and lipogenesis. Triglyceryl hydrolysis is attributed to generate free fatty acid by the anaerobic bacterium Propionibacterium acnes (P. acnes), a key role in inflammatory AV, reflects to the immune response which is stimulated via the toll-like receptor (TLR) 2 to Nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB) signaling pathway, thereafter induces the production of pro-inflammatory cytokines, chemokines and adhesion molecules.

   Current therapies for none or slightly inflammatory AV mostly use topical retinoids, moderate or severe acne use topical/oral antibiotics and oral isotretinoin. Topical antibiotics including clindamycin, erythromycin, nadifloxacin and tetracycline, are sometimes used in monotherapy but are more effective in combination with topical retinoids. For additional therapy, benzoyl peroxide, azelaic acid and sodium sulfacetamide, are antiseptic agent can use in combination treatment to decrease the risk of bacterial resistance. Severe acne uses oral antibiotics doxycycline, minocycline, tetracycline, erythromycin, and Trimethoprim/sulfamethoxazole combine topical treatment. Isotretinoin contributes to treat inflammatory papules, pustules and nodules, but it has been reported that isotretinoin has adverse effects teratogenic action in pregnant patients.

   More recently, clascoterone, an antiandrogen chemical had been shown efficacy in acne treatment.

   1.2 Introduction to investigational treatment(s) and other study treatment(s) 1.2.1 Overview of minoxidil Minoxidil was first used in anti-hypertension in clinical therapy. However, further study found minoxidil had the side effect of hirsutism, an abnormal hair growth over human body. Androgenetic alopecia (AGA) is an androgen-AR pathway may lead to hair loss, most frequent in men. In current clinical therapy, topical 2% or 5% solution of minoxidil have been used for AGA treatment but the therapeutic mechanism of minoxidil working on AGA is uncertain. The previous study showed minoxidil could reduce AR expression in messenger ribonucleic acid (mRNA) and protein level in Human Hair Dermal Papilla Cells (HHDPCs). Furthermore, the investigators demonstrated minoxidil could bind to AR protein structure at α8 and α11 helices which may hinder the association of interacting proteins, therefore disrupting downstream regulation of AR transactivation.
2. Study rationale:

   In the investigator's preliminary data, minoxidil could suppress fatty acid synthase activity and lipid formation in androgen-sensitive prostate cancer cell line in vitro. Minoxidil suppressed sebum formation in hamster flank organ in vivo. For P. acnes, minoxidil had a minimal inhibitory concentration of 5mM which was lower than 2% minoxidil (about 100mM). Furthermore, 2% and 5% minoxidil could suppress P. acnes induced infection/inflammation in animal studies. For acne formation, minoxidil could reduce sebum secretion, bacterial activity, and inflammation.
3. Study period (estimated):

   January, 2023~December, 2023
4. Objectives:

   4.1. primary: to test the toxicity of topical minoxidil in treatment of acne vulgaris.

   4.2. second: to evaluate the response and disease control rate in this pilot study.

   Measurement: Time to resolution of individual acne lesions (14 days) Split-face investigator's static global assessment (0, 1, 2, 4 wks) Acne lesion counts (0, 1, 2, 4 wks)
5. Methodology:

   This is a single institute, Division of Hemato-Oncology, Department of Internal Medicine and Department of Dermatology, Chang Gung Memorial Hospital, Linkou, Taiwan, randomized clinical trial.
6. Number of patients:

   Total 26 patients are needed and 13 patients for each group, 2% or 5% topical minoxidil solution treatment.
7. Diagnosis and main inclusion criteria:

7.1. Inclusion criteria:

1. Gender: both
2. Age limit: 20~50 year/old
3. Acne vulgaris: mild to moderate degree (Investigator's Global Assessment Scale:2~3)

7.2. Exclusion criteria: (1) pregnant or breast feeding woman (2) allergic to minoxidil or any ingredient of minoxidil solution including alcohol and propylene glycol (3) deny to discontinue topical therapy of acne more than 7 days before starting treatment (4) deny to discontinue systemic therapy of acne more than 28 days before starting treatment (5) alopecia under or ever using minoxidil, known androgen-AR pathway blocker (6) using shampoo containing minoxidil component in 28 days before starting treatment (7) irregular menstruation of known case of polycystic ovarian syndrome (8) Have had a facial procedure 2 weeks before the study start (9) using any oral contraceptives that have a specific anti-androgenic action 12 weeks before the study start

7.3. Accept Healthy Volunteers: No

8. Test products, dosage, mode of administration, and duration of treatment:

8.1. Minoxidil regimen: Panion & BF Biotech Inc. (PBF) Minoxidil Solution 5% Panion & BF Biotech Inc. (PBF) Minoxidil Solution 2%

8.2. Dosage

1. Minoxidil solution, 2% or 5%, topical, external, bid, D1~D14.
2. The daily applied amount must not exceed 2 ml.

8.3 Mode of administration

1. Two dosage of topical minoxidil will be tested, 2% and 5%.
2. Split face: 2% or 5% topical minoxidil solution applied and no treatment Description: Subjects will apply the 2% or 5% topical minoxidil solution to every inflammatory acne facial lesion on one half of the face and no treatment to every inflammatory acne lesion on the other half of the face twice a day for 4 weeks.

   *Split face mode: the investigators can't find support of the tested drug and placebo solution from Good Manufacturing Practice (GMP) factory in Taiwan. The investigators will use the patient's untreated half side of the face as control.
3. Monitor of treatment efficacy: number of inflammatory acne lesions counting, time to resolution of individual acne lesion, and degree of acne severity measurement.

   * (a) The enrolled patient will take 3 photos (left, right, and front) by using cell phone by the patient and send back to monitor center every night, day 0~ day 14. The treated side of face will be labeled.
   * (b) The enrolled patient will visit DERMA OPD on day1, 8, 15, and 29 and take photos.

8.4. duration of treatment This treatment cycle will be 14 days. Open label, randomization.

8.5. Concomitant treatment 8.5.1. Prohibited:

1. Any topical therapy of acne
2. Any systemic therapy of acne
3. Any medication, cosmetic products, or shampoo containing minoxidil component known androgen-AR pathway blocker
4. Any oral contraceptives that have a specific anti-androgenic action

9. Patient examination and re-evaluation:

1. Routine body temperature, and blood pressure, and pulse rate (TPR), and respiratory and body weight will be checked for screening and after treatment on day 8, 15, and 29.
2. Lab data of Complete Blood cell Count and Differential Count. (CBC/DC), creatinine, and Alanine Aminotransferase (ALT) will be checked for screening and routine checked after treatment on day 8, 15, and 29.
3. Minoxidil concentration measurement:

   * Serum minoxidil concentration will be checked before and after treatment 4hrs on day1, 24hrs on day2, on day8, and 15.
   * Urine minoxidil concentration will be checked on day2, 8, and 15.
4. Take photos:

   * (a) The enrolled patient will take 3 photos (left, right, and front) by using cell phone of the patient and send back to monitor center every night, day 0~ day 14. The treated side of the face will be labeled.
   * (b) The enrolled patient will take photos as baseline and visit DERMA OPD on day 8, 15, and 29 and take photos.

     10. Adverse events management, patient withdrawal criteria and study termination criteria When expected or unexpected adverse events (AEs) happened according to Worst Toxicity CTCAE v4.03 Grade, all will use the Hospital Information System (HIS) in Chang Gung Memorial Hospital (CGMH) to complete online notification within 24 hours after the physician or investigators informed. All these adverse events will be followed until to symptoms resolution/stable. These AEs data documents will be attached to interim and final report delivered to CGMH Institutional Review Board (IRB) and TFDA for integration. If expected or unexpected severe adverse events (SAEs) happened, all will not only complete online notification but also deliver the paper documents for CGMH IRB and Taiwan Food and Drug Administration (TFDA) within 24 hours after the physician or investigators informed.

Patients may continue treatment until they experience unacceptable toxicity that precludes any further treatment, until disease progression, and/or until treatment is discontinued at the discretion of the Investigator or by patient refusal.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: both
2. Age limit: 20~50 year/old
3. Acne vulgaris: mild to moderate degree (Investigator's Global Assessment Scale:2~3)

Exclusion Criteria:

1. pregnant or breast feeding woman
2. allergic to minoxidil or any ingredient of minoxidil solution including alcohol and propylene glycol
3. deny to discontinue topical therapy of acne more than 7 days before starting treatment
4. deny to discontinue systemic therapy of acne more than 28 days before starting treatment
5. alopecia under or ever using minoxidil, known androgen-AR pathway blocker
6. using shampoo containing minoxidil component in 28 days before starting treatment
7. irregular menstruation of known case of polycystic ovarian syndrome
8. Have had a facial procedure 2 weeks before the study start
9. using any oral contraceptives that have a specific anti-androgenic action 12 weeks before the study start

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure | Time to resolution of individual acne lesions (14 days)
  to test the toxicity of topical minoxidil in treatment of acne vulgaris.

SECONDARY OUTCOMES:
to evaluate the response of acne treatment in this pilot study. | Time to resolution of individual acne lesions (14 days)
  Take photos: acne numbers count changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Lung Hsu, Profesor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan